CLINICAL TRIAL: NCT01512056
Title: Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine,Formulation 2011-2012, in Dialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR-100-086
Record Dates: First submitted 2011-11-01; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: Influenza vaccine; dialysis; vaccine; Seroprotection; Seroresponse; Seroconversion; Safety of the vaccine
MeSH Terms: conditions — Influenza, Human; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the immunogenicity profiles of the AdimFlu-S (Experimental): Experimental group: to receive either only one dose of influenza vaccine at day 0 or one more booster vaccination 3 weeks later.
  Negative control group: dialysis patients who refused to receive influenza vaccination.
  Interventions: Drug: AdimFlu-S
- The safety outcome of the vaccine (No Intervention): Any adverse effect, including systemic or local site, will be recorded during the study period.

INTERVENTIONS:
Drug: AdimFlu-S — All enrolled participants will be divided into 3 groups: participants refused to receive vaccination, those receive either one (week 0) or one more booster vaccination (week 0 and week 3). Each dose of vaccine contains 15μg antigen of each virus strain suggested by WHO (A/California/7/2009 (H1N1);A/Perth/16/2009 (H3N2);B/Brisbane/60/2008).
  Arms: the immunogenicity profiles of the AdimFlu-S

SUMMARY:
The purpose of this study is to evaluate the antibody response in dialysis patents to each of the three influenza vaccine strains included in the licensed seasonal flu vaccine (Formulation 2011-2012).

DETAILED DESCRIPTION:
The immune response to influenza vaccine was poor in dialysis population than general population. The investigators want to evaluate another booster vaccination can improve the immune response in dialysis population. All enrolled participants will be divided into 3 groups: participants refused to receive vaccination, those receive either one (week 0) or one more booster vaccination (week 0 and week 3). The investigators will collect serum of participants 3 weeks, 6 weeks, 9 weeks and 18 weeks post vaccination and evaluate the difference of immune response in these 3 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females and aged more than 18 years;
2. Willing and able to adhere to visit schedules and all study requirements;
3. Subjects read and signed the study-specific informed consent.

Exclusion Criteria:

1. Subject or his/her family is employed by the participated hospital;
2. Subjects received 2010-2011 seasonal influenza vaccine within the previous 6 months;
3. History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication;
4. Personal or family history of Guillain-Barré Syndrome;
5. An acute febrile illness within 1 week prior to vaccination;
6. Current upper respiratory illness, including the common cold or nasal congestion within 72 hours;
7. Subjects with influenza-like illness as defined by the presence of fever (temperature ≥ 38°C) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
8. Female subjects who are pregnant during the study.
9. Patients who receive hemodialysis therapy less than 3 months.
10. Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
11. Immunodeficiency, or under immunosuppressive treatment.
12. Receipt of any vaccine within 1 week prior to study vaccination or expected receipt between Visit 1 (study vaccination) and Visit 2 (final collection of blood samples);
13. Receipt of any blood products, including immunoglobulin in the prior 3 months;
14. Any severe illness needed to be hospitalization within three months.
15. Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change of antibody titer before and after influenza vaccination | 18 weeks
  The primary endpoint will be the seroprotection rate which is defined as the proportion of subjects with HI titer ≥ 1:40. MicroNT-ELISA assay will also be used to evaluate the immune response post vaccination. The immune response based on microNT-ELISA antibody titers would be reported as antibody titer ≥1: 40 or ≥ 1:160 respectively because no threshold of protective NT antibody titer is clearly defined by the international guidelines.

SECONDARY OUTCOMES:
Seroresponse rate | 0, 3 weeks, 6 weeks, 9 weeks and 18 weeks
  The seroconversion is defined as the HI titer of the post-vaccination serum is at least 1:40 for those who had a negative pre-vaccination HI serum titer or a four-fold or greater increase in HI titers in subjects who had a positive pre-vaccination HAI serum titer.
Seroresponse rate | 0, 3 weeks, 6 weeks, 9 weeks and 18 weeks
  The seroresponse is defined as HI or micro-NT titer of the post-vaccination serum is at least 4-fold increase of the HI or micro-NT titer after vaccination.
  Geometric mean folds increase in HI or micro-NT titer.
the safety and tolerability profiles of the vaccine | 0, 3 week, 6 weeks, 9 weeks, 18 weeks
  evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of the AdimFlu-S manufactured by Adimmune Corporation.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan